CLINICAL TRIAL: NCT01084746
Title: Tailored Interactive Intervention to Increase CRCS
Acronym: PCCaSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sally Vernon, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SPH-01-084; R01CA097263-05 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal Cancer Screening; Computer Interactive Intervention; Predictors; Cost Effective Analysis; Transtheoretical Model

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PC-based tailored intervention (Active Comparator)
  Interventions: Behavioral: PC-based tailored intervention
- Printed educational materials (Active Comparator)
  Interventions: Behavioral: Printed educational materials
- No patient intervention (No Intervention): Patients will not receive a patient-directed intervention.

INTERVENTIONS:
Behavioral: PC-based tailored intervention — Patients will receive a tailored interactive PC-based intervention at a freestanding kiosk.
  Arms: PC-based tailored intervention
Behavioral: Printed educational materials — Patients will receive generic printed educational materials about CRCS in the PEC when they arrive at the Main Campus for their appointment.
  Arms: Printed educational materials

SUMMARY:
The primary goal of this research project is to conduct a 5-year prospective randomized trial of a theory-based intervention to increase patient completion of colorectal cancer screening (CRCS) among patients ages 50 to 64 years old.

DETAILED DESCRIPTION:
Specific Aim 1: Identify behavioral, social, and environmental factors associated with CRCS in male and female patients ages 50 to 64 years old in a primary care practice in Houston, Texas.

1.1. Update literature reviews of CRCS adherence. 1.2. Conduct secondary analysis of relevant data from other projects. 1.3. Conduct focus groups with primary care patients to determine their knowledge, attitudes, and beliefs about CRCS and to gather data to use for development of the educational intervention.

Specific Aim 2: Develop a personal computer (PC)-based tailored interactive intervention based on the transtheoretical (stages of change) model to increase CRCS in accordance with American Cancer Society (ACS) CRCS guidelines.

Specific Aim 3: Evaluate the effectiveness of the PC-based tailored interactive intervention for increasing CRCS through a randomized controlled trial.

Specific Aim 4: Analyze the relationship between a number of predictor variables and CRCS completion in order to develop a more complete conceptual framework for understanding screening adherence.

Specific Aim 5: Conduct a cost-effectiveness analysis of the PC-based tailored interactive intervention for increasing CRCS in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Receive primary care at the KSC Main Campus in Houston, Texas.
* Must have been patients at KSC for at least one year prior to enrollment in the study
* Be 50 to 64 years of age
* Have had CRC or adenomatous polyps
* Must agree to schedule a routine physical examination with their primary care provider and to complete a baseline interview

Exclusion Criteria:

-Have never been screened or be due for CRCS according to the ACS guidelines

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1224 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Increase patient completion of colorectal cancer screening (CRCS) among patients ages 50 to 64 years old. | 6months, 12months, 24 months
  6, 12, and 24 months post intervention, medical charts were reviewed to validate self-reported CRCS behavior.

SECONDARY OUTCOMES:
Secondary goals are to increase understanding of factors that predict completion of CRCS and to assess the cost-effectiveness of the intervention. | 6 months, 12 months, 24 months
  Survey data were collected at 6,12,and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sally W Vernon, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston School of Public Health, Houston, Texas, United States

REFERENCES:
- [Result] McQueen A, Tiro JA, Vernon SW. Construct validity and invariance of four factors associated with colorectal cancer screening across gender, race, and prior screening. Cancer Epidemiol Biomarkers Prev. 2008 Sep;17(9):2231-7. doi: 10.1158/1055-9965.EPI-08-0176. PMID 18768488
- [Result] Greisinger A, Hawley ST, Bettencourt JL, Perz CA, Vernon SW. Primary care patients' understanding of colorectal cancer screening. Cancer Detect Prev. 2006;30(1):67-74. doi: 10.1016/j.cdp.2005.10.001. Epub 2006 Feb 2. PMID 16458449
- [Result] Lairson DR, Chang YC, Bettencourt JL, Vernon SW, Greisinger A. Estimating development cost for a tailored interactive computer program to enhance colorectal cancer screening compliance. J Am Med Inform Assoc. 2006 Sep-Oct;13(5):476-84. doi: 10.1197/jamia.M2067. Epub 2006 Jun 23. PMID 16799126